CLINICAL TRIAL: NCT03743142
Title: Assessment of the GORE® EXCLUDER® Conformable AAA Endoprosthesis In the Treatment of Abdominal Aortic Aneurysms
Acronym: EXCeL
Status: Active, not recruiting | Type: Observational
Sponsor: Marc van Sambeek (Other)
Responsible Party: Sponsor-Investigator, Marc van Sambeek, prof. dr. M.R.H.M. van Sambeek, vascular surgeon, Catharina Ziekenhuis Eindhoven
Organization: Catharina Ziekenhuis Eindhoven (Other)
Other Study IDs: EXCeL
Record Dates: First submitted 2018-10-05; First posted 2018-11-16 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Abdominal Aortic Aneurysm (AAA)
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with AAA: Patients with AAA are eligible for participation and study screening. They will receive, once included, an endovascular repair of the AAA
  Interventions: Procedure: endovascular repair of the AAA

INTERVENTIONS:
Procedure: endovascular repair of the AAA — The Investigator will ensure that investigational devices are used only in subjects properly enrolled in the clinical study in accordance with the protocol. Subjects will undergo endovascular repair of their AAA. Procedural details may vary between sites, but will follow standard hospital protocol for EVAR and patient care management.

SUMMARY:
EVAR continues to evolve as a treatment option for AAA. New devices which are specifically designed to perform adequately across the spectrum of potential anatomic presentations for infrarenal EVAR are needed. The Department of Vascular Surgery at Catharina Hospital Eindhoven, The Netherlands initiates the EXCeL Registry.

This study will assess the safety and effectiveness of the GORE® EXCLUDER® Conformable AAA Endoprosthesis (CEXC Device) in patients who meet the IFU anatomic criteria (≥15mm proximal neck length and ≤90˚ proximal neck angulation; and ≥10mm proximal neck length and ≤60˚ proximal neck angulation) and in patients with challenging anatomic presentation that may present outside the IFU anatomic criteria. Successful outcomes from this study will provide evidence to support the CEXC Device as an option for expanding EVAR to a broader patient population with more challenging anatomic presentations.

DETAILED DESCRIPTION:
EXCeL Registry is a multi-center, post-market, non-interventional, non-randomized, single-arm, prospective observational study, initiated by the Department of Vascular Surgery at Catharina Hospital Eindhoven, The Netherlands. The study has a single-arm without controls, as it is descriptive in nature, 150 consented subjects from up to 10 high-volume sites across Europe will be included into this registry.

Study enrollment is open to consecutively enrolled subjects who in the opinion of the investigator and according to Table A (p.9) -Anatomic measurement table and group specific- are suitable for being treated. An independent core lab will validate pre-requisite anatomy measurement to evaluate candidates for endovascular AAA repair with the GORE® EXCLUDER® Conformable AAA Endoprosthesis.

EXCeL Registry does not intervene with the physician's decision to choose for endovascular treatment with a GORE® EXCLUDER® Conformable AAA Endoprosthesis. Follow-up measurements are requested at 1 month, 12 months, and yearly thereafter, as minimally required by the reporting standards for endovascular aortic aneurysm repair. Beyond this, sites can schedule the subject's follow-up visits as usual in their clinical practice, as this study does not intervene in or influence the follow-up regimen. For data completion it is, however, possible that a telephone-contact with subjects will be requested.

This study will assess the safety and effectiveness of the GORE® EXCLUDER® Conformable AAA Endoprosthesis in patients who meet the IFU anatomic criteria and in patients with challenging anatomic presentation that may fall outside the IFU anatomic criteria and identified in the protocol as challenging anatomy treatment cohort. Consented subjects placed in the challenging anatomy cohort will be followed per the protocol and any data analysis on this cohort will be descriptive in nature only.

Up to 11 clinical investigative Sites will enroll a total of 150 subjects to allow for the broad range of aortic necks lengths and aortic neck angulations to be in the study. Consecutive consented subjects meeting protocol criteria will be part of the enrollment strategy:

* Subjects with neck length of ≥15 mm and neck angulation of ≤90°
* Subjects with neck length of ≥10 mm and neck angulation of ≤60˚ An independent Core Lab will read each subjects' pre-operative CT images and measure neck length and neck angle. These core lab measurements will determine if subject's anatomy meets IFU criteria (regarding neck length and neck angle) or if this subject has to be placed in the challenging anatomy treatment cohort.

The EXCeL Registry, by itself, has a prospective observational study design, and focuses on patients with infrarenal abdominal or aorto-iliac aneurysms with Regular and challenging anatomy, scheduled for EVAR treatment with the GORE® EXCLUDER® Conformable AAA Endoprosthesis. No hypotheses testing will be carried out within this study design. However, the EXCeL Registry aims at creating a database that can analyze the performance of the GORE® EXCLUDER® Conformable AAA Endoprosthesis in different anatomies.

Sample size calculation was precision based in order to achieve a desirable confidence interval width. An assumption of freedom from any endpoint event of 90% and a desired Confidence Interval (CI) of 10% or less results in a sample size of 150. Calculations performed with PASS13.

A Subject will be considered lost to follow-up and withdrawn from the study once they have missed two consecutive follow-up visits and three documented attempts have been made by the Investigator or designee to contact the Subject or next of kin. In the event that the Subject is lost to follow-up, the date of discontinuation of the study will be recorded as the last contact with the Subject by the investigative site.

A Subject has completed the study when they have completed the three year follow-up visit. Any Subject that does not complete these requirements due to voluntary withdrawal, physician withdrawal, death, or any other reason will be considered a withdrawal.

Data collected on each subject will be recorded on an online electronic CRF. A paper version of the CRFs may be printed at the sites to use as a working copy. Instructions for proper completion of the electronic CRF and how to use it online will be provided to the clinical site. The investigator or an authorized member of the investigational team must sign all completed CRFs, by using a unique signature code. This code will be provided to the user at the start of the study.

The Statistics & Data Analysis team at the Department of Vascular Surgery, Catharina Hospital, Eindhoven will check the data entered on the CRFs for consistency and completeness on a regular basis, both manually as well as by using statistical monitoring of the clinical database. Sites will be contacted for data inconsistencies in order to recover incomplete, inconsistent, or missing data.

In case of multiple futile attempts of data completeness data and non-respond from clinical sites monitors of the Department of Vascular Surgery, Catharina Hospital, Eindhoven will visit sites. They will then collect data from source documents in a final attempt to complete the applicable CRFs. To enhance data quality, additional site visits may be conducted to crosscheck CRFs with patient files in approximately 20% of enrolled subjects. The local investigator will timely be informed of this scheduled visit.

ELIGIBILITY:
Inclusion Criteria:

1. AAA meeting any of the following criteria:

* Maximum diameter ≥50 mm
* Rapid growth (>5 mm in a 6 month period)
* Non-ruptured AAA presenting with clinical symptoms 2 Adequate anatomy to receive the CEXC Device, including:
* Adequate iliac / femoral access
* Infrarenal aortic neck diameter 16-32 mm
* Distal iliac artery seal zone ≥10 mm
* Iliac artery diameter 8-25 mm 3. An Informed Consent Form (ICF) dated and signed by subject 4. Male or infertile female* 5. Able to comply with protocol requirements including following-up 6. Life expectancy >2 years 7. Age ≥18 years * Infertile female - condition which prevents pregnancy, e.g., hysterectomy, tubal ligation or post-menopausal for greater than 1 year

Exclusion Criteria:

1. Mycotic or ruptured aneurysm
2. Saccular aneurysm, unless it meets inclusion criteria of rapid growth (>5 mm in a 6 month period) or maximum diameter of (≥50 mm)
3. Known concomitant thoracic aortic aneurysm which requires surgical intervention 4. Renal insufficiency defined as creatinine >2.5 mg/dL or GFR <30 mL/min/1.73 m2

5. Patient has body habitus or other medical condition which prevents adequate delineation of the aorta 6. Participating in another investigational device study within 1 year of treatment 7. Systemic infection which may increase the risk of endovascular graft infection 8. Known degenerative connective tissue disease, e.g. Marfan or Ehler-Danlos Syndrome 9. Planned concomitant surgical procedure or major surgery within 30 days of treatment date, including planned branched, snorkel or chimney procedures 10. Known sensitivities or allergies to the device materials 11. Use of non-Gore stent grafts in initial procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AAA are eligible for participation and study screening.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Primary safety success defined by the absence of major adverse events | up to 30 days after index procedure
  These major adverse events are defined as all-cause mortality, stroke, mycardial infarction, bowel ischemia, paraplegia, respiratory failure, renal failure and thromboembolic events (including limb occlusion and distal embolic events).
Technical treatment success | At the primary procedure
  Proportion of subjects who experience successful, delivery and deployment of all required EXCC Device components annd successful removal of EXCC device delivery catheter(s)
Clinical effectiveness success | From the day after the initial procedure up to 3 years after the initial procedure (which is the end of the follow up period for this registry
  Effectiveness defined as absence of type I endoleak at each visit, Type III endoleak at the 12 month visit, migration (10 mm or more) between the one month and the 12 month visit, AAA enlargement >5 mm with or without intervention between the one month and the 12 month visit, AAA rupture through the 12 month visit, conversion to open repair through the 12 month visit, limb occlusion

SECONDARY OUTCOMES:
Incidence of treatment-emerged adverse events (safety) | From hospital admission before index procedure up to study completion after the 3 years follow up
  30 day major adverse events, individual elements of the primary safety and effectiveness endpoints, secondary procedures, type II endoleak, type IV endoleak, index procedure blood loss, index procedure time, length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: M.R.H.M. van Sambeek, Prof. dr., Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (8):
- APHP Hopital Européen, Paris, France
- San Martino Hospital, Genova, Italy
- Netherlands (3):
  - Rijnstate Hospital, Arnhem
  - Catharina Hospital, Eindhoven
  - ETZ, Tilburg
- Spain (2):
  - San Carlos Hospital, Madrid
  - Complexo Hospitalario de Orense, Ourense
- North Bristol NHS Trust, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data collected on each subject will be recorded on an online electronic CRF. A paper version of the CRFs may be printed at the sites to use as a working copy. Instructions for proper completion of the electronic CRF and how to use it online will be provided to the clinical site. The investigator or an authorized member of the investigational team must sign all completed CRFs, by using a unique signature code. This code will be provided to the user at the start of the study.
  All records and other information about subjects participating in this registry will be treated as confidential. The sponsor, Department of Vascular Surgery, Catharina Hospital, Eindhoven, will collect data and monitors study records.Study data may be made available to third parties, e.g., in the case of an audit performed by regulatory authorities, provided the data are treated confidentially and that the subject's privacy is guaranteed.
Supporting Information: Study Protocol, ICF